CLINICAL TRIAL: NCT06047990
Title: Endobiliary Percutaneous Cryobiopsy in Malignant Biliary Obstruction
Acronym: BICRYOB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Tomas Andrasina, Tomáš Andrašina, MD, PhD; Assistant professor, Head of Non-vascular interventions and Computed Tomography of the Department of Radiology and Nuclear Medicine, Brno University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: FNBKRNM0003
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Biliary Tract Carcinoma; Biliary Obstruction
Keywords: cryobiopsy; biliary obstruction; percutaneous transhepatic drainage

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomization was performed by the Institute of Biostatistics and Analysis of Masaryk University Brno.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryobiopsy (Experimental): In randomised patients in experimental arm was initially performed cryobiopsy (3 samples) and cosequently forceps biopsy (6 samples) with 5.2F or 7.5F forceps. Both sampling techniques were performed during one procedure of percutaneous transhepatic drainage under fluoroscopic control.
  Interventions: Device: Cryobiopsy catheter
- Forceps biopsy (Active Comparator): In randomised patients in control arm was initially performed forceps biopsy (6 samples) with 5.2F or 7.5F forceps and cosequently cryobiopsy (3 samples). Both sampling techniques were performed during one procedure of percutaneous transhepatic drainage under fluoroscopic control.
  Interventions: Device: Cryobiopsy catheter

INTERVENTIONS:
Device: Cryobiopsy catheter — Comparison of endobiliary forceps biopsy and cryobiopsy of biliary stenosis during percutaneous transhepatic drainage.

SUMMARY:
The rationale of the study is to explore the safety and efficacy of percutaneously performed endobiliary cryobiopsy in patiens with histologically unverified biliary stenosis.

DETAILED DESCRIPTION:
In patients with malignant biliary stenosis in whom endoscopic retrograde cholangiography (ERCP) is not feasible , percutaneous transhepatic drainage (PTD) is indicated. Biopsy is required for further management of the patient. In patients unsuitable for biopsy under CT or endoscopic guidance, samples can be collected endobiliary by PTD. The biopsy vie PTD can be sampled either at the initial drainage using disposable 5.2F forceps or delayed after 2 or more days using 7.5F endobiliary forceps. An alternative to this procedure is endobiliary sampling by cryobiopsy using 1.1mm, 1.7mm or 2.4mm catheters. To minimize bias, each patient will be sampled both by cryobiopsy and forceps biopsy. The order of cryobiopsy and forceps biopsy will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* biliary stenosis of unknown etiology
* unsuccessful or unfeasable ERCP
* indicated percutaneous transhepatic drainage

Exclusion Criteria:

* histologically verified biliary stenosis
* INR ≥ 1,5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of biopsy sampling to detect malignancy | up to month 12 or death of the patient
  Comparison of sensitivity of endobiliary cryobiopsy and forceps biopsy for detection of malignancy.
Quality of samples collected by endobiliary cryobiopsy and forceps biopsy - weight | up to month 12 or death of the patient
  Comparison of weight (in milligrams) of samples collected by endobiliary cryopsy and forceps biopsy. Each sample will be weighed separately and one measurement value will be recorded for each sample.
Quality of samples collected by endobiliary cryobiopsy and forceps biopsy - size | up to month 12 or death of the patient
  Comparison of the size weight (in millimeters) of samples collected by endobiliary cryopsy and forceps biopsy. Each sample will be weighed in two dimensions on slide.

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No